CLINICAL TRIAL: NCT02098434
Title: Implication of Ovarian Hormones in the Neural Correlates of Stress Induced Drug Craving
Brief Title: Ovarian Hormones and Stress Induced Drug Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19884
Record Dates: First submitted 2012-10-22; First posted 2014-03-28 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2014-11

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Montreal Imaging Stress Task (Experimental): Math task to induce stress response
  Interventions: Behavioral: Montreal Imaging Stress Task

INTERVENTIONS:
Behavioral: Montreal Imaging Stress Task — Math task developed to induce a stress response in a laboratory setting
  Other Names: MIST

SUMMARY:
The study is investigating the impact of progesterone and estrogen on brain areas that are involved with stress response and drug craving. The study will involve 40 women who will participate in the Montreal Imaging Stress Task (MIST) while undergoing fMRI scanning procedures. Half of the women will complete the procedures during the luteal phase of the menstrual cycle; the other half will complete procedures during the follicular phase. Subjective and physiological measures (cortisol levels) will be used to measure stress and craving response. Hypothesis 1A is that all women will exhibit increased craving, stress response, salivary cortisol and BNST and limbic nuclei activation in response to the MIST task. Hypothesis 1B is that these increased responses will be higher for women in the luteal phase than for women in the follicular phase of the menstrual cycle.

ELIGIBILITY:
GGeneral Inclusion / Exclusion Criteria Inclusion Criteria

1. Pre-menopausal. Individuals who are no longer menstruating regularly will not be included as we are examining ovarian hormone status on stress reactivity.
2. Right-handed
3. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
4. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for a three-day period immediately prior to the CTRC admission. Participants must have a negative breathalyzer, urine drug screen.
5. Subjects must consent to outpatient admission to the CTRC.

Exclusion Criteria

1. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect HPA axis function.
2. Subjects with any liver function test of greater than two times normal, as compromised liver function can interfere with HPA axis activity.
3. Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect HPA axis function.
4. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with HPA function.
5. Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents, that interfere with HPA axis function within one month of the time of testing.
6. Subjects taking opiates, opiate antagonists, or benzodiazepines. (Subjects who have been maintained on SSRI's, anticonvulsants, or antipsychotics (for sleep only) for more than 8 weeks or longer are NOT excluded).
7. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
8. Subjects with any acute illness or fever as this may affect HPA axis activity. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
9. Subjects who are > 30% over ideal weight or have a BMI greater than 35 will be considered for study participation based on the clinical judgment of study staff.
10. Subjects who are unwilling to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for three days prior to the stress task procedure.
11. Persons with ferrous metal implants or pacemaker since fMRI will be used.
12. Subjects that are claustrophobic.
13. Males.
14. Women taking birth control pills, or Depo Provera (medroxyprogesterone acetate).

Inclusion Criteria Cocaine-Dependent Women a. Women meeting criteria for cocaine-dependence in the previous three months (current).

Exclusion Criteria Cocaine-Dependent Women

a. Subjects meeting DSM-IV criteria for current dependence (within 2 months) on substances other than cocaine. Nicotine dependence can affect HPA function therefore it would be ideal to exclude subjects with nicotine use. Because of the comorbidity of cocaine and nicotine dependence, this would seriously compromise the feasibility of recruitment. Alcohol has also been known to affect HPA function, however to enhance recruitment efforts, individuals with alcohol dependence or abuse will be included in the study if they do not require medically supervised detoxification.

Inclusion Criteria Non-Dependent Healthy Control Women a. As above. Exclusion Criteria Non-Dependent Healthy Control Women

a. Women meeting DSM-IV criteria for past or current substance dependence (other than nicotine).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD)signal activation in limbic brain regions | Scan visit, before and after MIST (day 1)
  Exposure to the MIST task will increase activation in these brain areas as measured by fMRI scanning procedures, and the increase will be more pronounced for women in the luteal rather than follicular phase of the menstrual cycle.

SECONDARY OUTCOMES:
Stress response on 0-10 Likert scale | Scan visit, before and after MIST (day 1)
  Participants are asked to rate stress on a 10-point Likert scale. It is hypothesized that subjective ratings will increase following the MIST task, and that the increase will be more pronounced for women in the luteal rather than follicular phase of the menstrual cycle.
Subjective craving on 0-10 Likert scale | Scan visit, before and after MIST (day 1)
  Participants are asked to rate craving on a 10-point Likert scale. It is hypothesized that craving greater after completion of the MIST than before the MIST task, and that the increase will be more pronounced for women in the luteal rather than follicular phase of the menstrual cycle.

OTHER OUTCOMES:
Salivary cortisol levels | Scan visit, before and after MIST (day 1)
  Salivary samples will be collected throughout scanning procedures to determine salivary cortisol levels. It is hypothesized that cortisol levels will increase following the MIST task, and that the increase will be more pronounced for women in the luteal rather than follicular phase of the menstrual cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States